CLINICAL TRIAL: NCT04418232
Title: Feasibility of a Novel Systems Approach for Improving Utilization of Alzheimer's Disease Services Among Latinos Attending Primary Care Practices
Brief Title: Feasibility of a Systems Approach for Alzheimer's Services Among Latinos Attending Primary Care Practices
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00145615
Record Dates: First submitted 2020-06-02; First posted 2020-06-05 (Actual); Results first posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Alianza Latina (Experimental): The main components of Alianza Latina are 1) providing primary care providers with education, training and tools for timely dementia diagnosis and optimal treatment and 2) providing Latino dementia patients with enhanced chronic care through bilingual Health Navigators.
  Interventions: Combination Product: Alianza Latina

INTERVENTIONS:
Combination Product: Alianza Latina — The main components of Alianza Latina are 1) providing primary care providers with education, training and tools for timely dementia diagnosis and optimal treatment and 2) providing Latino dementia patients with enhanced chronic care through bilingual Health Navigators.

SUMMARY:
The research team will train primary care practitioners from Kansas City clinics to enhance skills in cultural competence, dementia detection, treatment and referral to a Health Navigator among Latinos 65 and older with dementia. The Health Navigator will provide patient/caregiver dyads referred by Alianza Latina providers with care management, psychosocial support and links to relevant community resources. Outcomes include feasibility and acceptability of 1) PCP training and 2) patient and caregiver dementia care.

DETAILED DESCRIPTION:
Alzheimer's disease and related dementias (ADRD) are a major cause of mortality and disability in later life and cost the US healthcare system more than cancer or heart disease. The National Alzheimer's Plan Act and the National Institutes of Health have identified ADRD disparities among ethnic minorities as a public health priority. Latinos with ADRD experience substantial disparities with reduced rates of early diagnosis and lower quality care compared to their non-Latino white peers, which put them at an increased risk for steeper cognitive decline, morbidity, mortality and higher caregiver burden. A number of barriers conspire to create these disparities including a lack of an evidence-based strategy to address ADRD in clinics, patient and primary care provider (PCP) reduced ADRD knowledge, negative attitudes regarding ADRD, PCP's lack of time, cultural and language barriers and health insurance status. To improve healthcare delivery to Latinos with ADRD, researchers need to redesign current ADRD detection and care systems to follow evidence-based recommendations for early detection and culturally appropriate chronic care.

The overall aim of this proposal is to enhance the delivery of ADRD services to Latinos in primary care through a scalable systems approach that includes evidence-based recommendations. Primary care clinics are the ideal setting to provide ADRD services, as 93% of older Latinos have a usual source of healthcare. The novel systems approach (Alianza Latina/Latino Alliance) will enhance timely ADRD diagnosis and optimal care to minimize behavioral symptoms and cognitive decline among Latinos in a linguistically and culturally-appropriate way. Alianza Latina will use the Collaborative Care Framework that capitalizes on PCPs and Health Navigators. 1) PCPs will undergo evidence-based training to enhance timely and culturally appropriate diagnosis and implement it in their work routine. 2) PCPs will detect, treat and refer Latino ADRD patients to a bilingual Health Navigator to provide chronic care management, which will reduce PCP time burden.

Aim 2: Test the feasibility and acceptability of Alianza Latina. Aim 2.a: The research team will train PCPs from Kansas City clinics to enhance skills in cultural competence, ADRD detection, treatment and referral to a Health Navigator among Latinos 65 and older with ADRD. Aim 2.b. The Health Navigator will provide patients/caregiver dyads referred by Alianza Latina PCPs with care management, psychosocial support and links to relevant community resources. The research team will assess the feasibility and acceptability of 1) PCP training and 2) patient and caregiver ADRD care. Caregivers will be enrolled in a text messaging program, called CuidaTEXT, that will educate about memory and thinking problems, solve problems that are common among families with memory and thinking problems, send reminders for appointments and medications, and improve communication with the PCP, family, friends, and other resources.

ELIGIBILITY:
Inclusion Criteria for care recipients within the dyad:

* Identify as Latino
* Community dwelling
* Diagnosed with mild cognitive impairment or dementia
* Have a caregiver 18 years old or older
* Have co-participant with access to a privately-owned cell phone with a flat fee for text messages

Inclusion Criteria for primary care providers:

* Be 18 years old or older
* Work as a primary care provider in the US

Exclusion Criteria for care recipients within the dyad:

* Not identify as Latino
* Not community dwelling
* Not diagnosed with mild cognitive impairment or dementia
* Not having a caregiver 18 years old or older
* Not having a co-participant with access to a privately-owned cell phone with a flat fee for text messages

Exclusion Criteria for primary care providers:

* Younger than 18 years old
* Not work as a primary care provider in the US

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Perales Puchalt, PhD, MPH, Principal Investigator — KUMC
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
The final dataset will include patients' and caregivers' demographic and behavioral data from interviews as well as metrics and feasibility information provided by the primary care providers. Along with the dataset, we will create a code book documenting all variables. Study participants may find their diagnosis information potentially stigmatizing, and may prefer that these diagnoses remain entirely confidential. Although the data analytic files will not have direct identifiers (only study identification numbers), the possibility of deductive disclosure of subjects with certain clinical characteristics may remain. To safeguard against the unlikely event of deductive disclosure, we will only make the data files and codebook available to other researchers on a case-by-case basis.
Supporting Information: Study Protocol
Time Frame: February 1, 2025
Access Criteria: Researchers requesting data will need to complete a request form outlining intended use of the data, and agree to use the data solely for this intended purpose. Prior to data release, researchers requesting data will be required to sign a confidentiality agreement specifying that they will not identify any individual participant, that they will use secure technology to safeguard the data, and that they will destroy or return the data after their analyses are completed.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study includes 100 dyads. Each dyad is formed by a unique caregiver and a care recipient. Ten care recipients are in more than one dyad, as more than one of their caregivers participated in the study.
Groups:
- Alianza Latina: The main components of Alianza Latina were:
  1. Primary care provider education: This training was informed by the Health Belief Model and Social Learning Theory and included clinically-focused lectures, case examples with discussion, videos and materials. Topics included dementia detection and diagnosis, treatment, and care, early detection, patient empowerment, and cultural competence. The modality of all training events was live and online via videoconferences.
  2. Coordinated care: This program provided Latino dementia patients with enhanced chronic care through bilingual Health Navigators. Alianza Latina is a six-month bilingual intervention, designed to cater to the unique needs of Latino caregivers. It integrates CuidaTEXT, an SMS program, with monthly phone consultations facilitated by a trained coach from the research team. These consultations aim to identify unaddressed needs and provide necessary support. Participants in CuidaTEXT receive scheduled messages and can also request on-demand assistance by texting. CuidaTEXT entails sending 1-3 automated daily messages covering various aspects such as logistics, dementia education, self-care, social support, end-of-life care, managing dementia-related behaviors, and problem-solving strategies. Additionally, participants could text keyword-based queries for immediate assistance on the above-mentioned topics and engage in live chat sessions with the coach for further guidance upon request.
Period: Overall Study
Arm/Group | Alianza Latina
Started (This number includes 100 caregivers of 84 care recipients who underwent the Alianza Latina care support intervention; 26 caregivers were part of 10 clusters of 2 (n=5), 3 (n=4), and 4 (n=1) caregivers of the same person with dementia. This number also includes results from 59 primary care providers who underwent a dementia training delivered as standard training by the KU Alzheimer's Disease Research Center.) | 243
Completed (This number includes 88 caregivers of 73 care recipients who completed the Alianza Latina study. This number also includes results from 11 primary care providers who completed the 6-month survey after the dementia training delivered as standard training by the KU Alzheimer's Disease Research Center.) | 172
Not Completed | 71

BASELINE CHARACTERISTICS:
Population: Analyses include the 59 primary care providers from aim 2a, and the 100 caregivers and 84 care recipients that form the 100 dyads from Aim 2b. Each dyad is formed by a unique caregiver and a care recipient. Ten care recipients are in more than one dyad, as more than one of their caregivers participated in the study. For clarity of results, baseline variables refer to care recipients unless the variable name states that it refers to a different sample (caregiver or primary care provider).
Arm/Group | Alianza Latina
Number analyzed (Participants) | 243
Age, Categorical [Count of Participants; unit: Participants] — Population: Number analyzed in row differs from overall because we are reporting different samples (care recipients, caregivers and primary care providers).
  Participants
    Care recipients: number analyzed (Participants) | 84
    Care recipients: <=18 years | 0
    Care recipients: Between 18 and 65 years | 8
    Care recipients: >=65 years | 76
    Caregivers: number analyzed (Participants) | 100
    Caregivers: <=18 years | 0
    Caregivers: Between 18 and 65 years | 90
    Caregivers: >=65 years | 10
    Primary care providers: number analyzed (Participants) | 59
    Primary care providers: <=18 years | 0
    Primary care providers: Between 18 and 65 years | 47
    Primary care providers: >=65 years | 12
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Number analyzed in row differs from overall because we are reporting different samples (care recipients, caregivers and primary care providers)
  years
    Care recipients: number analyzed (Participants) | 84
    Care recipients | 78.2 (10.2)
    Caregivers: number analyzed (Participants) | 100
    Caregivers | 52.0 (10.2)
    Primary care providers: number analyzed (Participants) | 59
    Primary care providers | 49.5 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Number analyzed in row differs from overall because we are reporting different samples (care recipients, caregivers and primary care providers).
  Participants
    Care recipients: number analyzed (Participants) | 84
    Care recipients: Female | 71
    Care recipients: Male | 13
    Caregivers: number analyzed (Participants) | 100
    Caregivers: Female | 82
    Caregivers: Male | 18
    Primary care providers: number analyzed (Participants) | 59
    Primary care providers: Female | 42
    Primary care providers: Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Number analyzed in row differs from overall because we are reporting different samples (care recipients, caregivers and primary care providers).
  Participants
    Care recipients: number analyzed (Participants) | 84
    Care recipients: Hispanic or Latino | 84
    Care recipients: Not Hispanic or Latino | 0
    Care recipients: Unknown or Not Reported | 0
    Caregivers: number analyzed (Participants) | 100
    Caregivers: Hispanic or Latino | 95
    Caregivers: Not Hispanic or Latino | 4
    Caregivers: Unknown or Not Reported | 1
    Primary care providers: number analyzed (Participants) | 59
    Primary care providers: Hispanic or Latino | 3
    Primary care providers: Not Hispanic or Latino | 50
    Primary care providers: Unknown or Not Reported | 6
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Number analyzed in row differs from overall because we are reporting different samples (care recipients, caregivers and primary care providers).
  Participants
    Care recipients: number analyzed (Participants) | 84
    Care recipients: American Indian or Alaska Native | 0
    Care recipients: Asian | 0
    Care recipients: Native Hawaiian or Other Pacific Islander | 0
    Care recipients: Black or African American | 1
    Care recipients: White | 15
    Care recipients: More than one race | 0
    Care recipients: Unknown or Not Reported | 68
    Caregivers: number analyzed (Participants) | 100
    Caregivers: American Indian or Alaska Native | 0
    Caregivers: Asian | 0
    Caregivers: Native Hawaiian or Other Pacific Islander | 0
    Caregivers: Black or African American | 1
    Caregivers: White | 25
    Caregivers: More than one race | 2
    Caregivers: Unknown or Not Reported | 72
    Primary care providers: number analyzed (Participants) | 59
    Primary care providers: American Indian or Alaska Native | 4
    Primary care providers: Asian | 0
    Primary care providers: Native Hawaiian or Other Pacific Islander | 0
    Primary care providers: Black or African American | 2
    Primary care providers: White | 46
    Primary care providers: More than one race | 4
    Primary care providers: Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 243
Caregivers' relation to care recipients [Count of Participants; unit: Participants] — Population: Number analyzed in row differs from overall because it only refers to caregivers' relation to care recipients.
  Participants
    number analyzed (Participants) | 100
    Children | 73
    Partner | 11
    Children-in-law | 4
    Other | 12
Dementia diagnosis [Count of Participants; unit: Participants] — Population: Number analyzed in row differs from overall, because analyses only refer to care recipients.
  Participants
    number analyzed (Participants) | 84
    Alzheimer's dementia | 38
    Unspecified dementia | 27
    Vascular dementia | 5
    Lewy Bodies/Parkinson's dementia | 5
    Mixed dementia | 4
    Frontotemporal dementia | 2
    Other | 2
    Mild Cognitive Impairment | 1
Years of education [Mean (Standard Deviation); unit: years] — Population: Number analyzed in row differs from overall because we are reporting different samples (care recipients and caregivers).
  years
    Care recipients: number analyzed (Participants) | 84
    Care recipients | 11.2 (20.4)
    Caregivers: number analyzed (Participants) | 100
    Caregivers | 12.4 (4.4)

OUTCOME MEASURES:

1. Primary Outcome: Provider Recruitment Feasibility
Description: Metrics of the number of providers who agree to be trained per month
Time Frame: During the 9 months of the provider intervention period
Measure: Mean (Standard Deviation); unit: Providers trained per month
Arm/Group | Alianza Latina
Number analyzed (Participants) | 59
Providers trained per month | 1.44 (2.74)

2. Primary Outcome: Provider Retention Feasibility
Description: Metrics of the percentage of providers who continue to partner with the study team by the end of the provider intervention period
Time Frame: During the 9 months of the provider intervention period
Population: Primary care providers that are part of Aim 2a
Measure: Count of Participants; unit: Participants
Arm/Group | Alianza Latina
Number analyzed (Participants) | 59
Participants | 11

3. Primary Outcome: Provider Fidelity Feasibility 1
Description: Percentage of providers able to implement screenings in regular workflow, measured via survey with the question "To what extent were you able to implement screenings in regular workflow" with three response options: "not at all", "to some degree", "usually", "almost always" and "always"
Time Frame: 9 months (end of the provider intervention period)
Population: Primary care providers that are part of Aim 2a
Measure: Count of Participants; unit: Participants
Arm/Group | Alianza Latina
Number analyzed (Participants) | 59
Participants
  not at all | 1
  to some degree | 5
  usually | 19
  almost always | 9
  always | 8
  Missing | 17

4. Primary Outcome: Provider Assessment Feasibility 1
Description: Metrics of the percentage of providers who complete baseline and follow-up surveys about dementia knowledge, attitudes and skills
Time Frame: During the 9 months of the provider intervention period
Population: Primary care providers that are part of Aim 2a
Measure: Count of Participants; unit: Participants
Arm/Group | Alianza Latina
Number analyzed (Participants) | 59
Participants | 43

5. Primary Outcome: Provider Fidelity Feasibility 2
Description: Metrics of the Number of referrals to Health Navigator per month
Time Frame: During the 9 months of the provider intervention period
Population: Primary care providers that are part of Aim 2a
Measure: Mean (Standard Deviation); unit: Referrals per month
Arm/Group | Alianza Latina
Number analyzed (Participants) | 59
Referrals per month | 5.77 (3.45)

6. Primary Outcome: Overall Provider Satisfaction With Training
Description: Survey question including a 5-item Likert scale on satisfaction with training (not at all to very much)
Time Frame: 9 months (end of the provider intervention period)
Population: Primary care providers that are part of Aim 2a
Measure: Count of Participants; unit: Participants
Arm/Group | Alianza Latina
Number analyzed (Participants) | 59
Participants
  Not at all | 0
  Slightly | 2
  Moderately | 4
  very much | 15
  Extremely | 21
  Missing | 17

7. Primary Outcome: Importance of Navigators to Providers
Description: Survey question including a 5-item Likert scale on the perceived importance of Navigators to providers (not at all to very much)
Time Frame: 9 months (end of the provider intervention period)
Population: Primary care providers that are part of Aim 2a (Only among the people who reported using health navigators)
Measure: Count of Participants; unit: Participants
Arm/Group | Alianza Latina
Number analyzed (Participants) | 1
Participants
  Not at all | 0
  Slightly | 0
  Moderately | 0
  Very much | 0
  Extremely | 1

8. Primary Outcome: Participant Recruitment Fidelity
Description: Metrics of percentage of referred Latino dementia dyads who enroll in Health Navigator services
Time Frame: During the 15 months of the whole intervention period
Population: The Overall Number of Participants Analyzed is greater than the number Started in the Participant Flow because this variable reports the dyads who end up enrolling (100) out of the ones referred (127)
Measure: Number; unit: Percentage of dyads
Arm/Group | Alianza Latina
Number analyzed (Participants) | 127
Percentage of dyads | 78.7

9. Primary Outcome: Participant Retention Fidelity
Description: Metrics of percentage of referred Latino dementia dyads followed up at six months
Time Frame: During the 6 months of the Navigator intervention period
Population: The Overall Number of Participants Analyzed is greater than the number Started in the Participant Flow because this variable reports the dyads who are followed up (88) out of the ones referred (127)
Measure: Number; unit: Percentage of dyads
Arm/Group | Alianza Latina
Number analyzed (Participants) | 127
Percentage of dyads | 69.3

10. Primary Outcome: Participant Assessment Fidelity
Description: Metrics of the percentage of planned baseline and follow-up survey ratings completed
Time Frame: During the 6 months of the Navigator intervention period
Population: Participants responding to these are dyads (caregivers and, when possible, care recipients)
Measure: Number; unit: Percent of dyads
Arm/Group | Alianza Latina
Number analyzed (Participants) | 100
Percent of dyads | 77

11. Primary Outcome: Participant Treatment Adherence
Description: Metrics of the percentage of referred Latino dementia dyads who attend at least 50% of Health Navigator visits
Time Frame: During the 6 months of the Navigator intervention period
Population: Participants responding to these are dyads (caregivers and, when possible, care recipients)
Measure: Number; unit: Percentage of dyads
Arm/Group | Alianza Latina
Number analyzed (Participants) | 100
Percentage of dyads | 29

12. Primary Outcome: Overall Participant Satisfaction With the Clinic Side of the Intervention
Description: Survey question including a 5-item Likert scale on caregivers' satisfaction with clinic services (not at all to very much)
Time Frame: 6 months after baseline
Population: Participants responding to these are caregivers
Measure: Count of Participants; unit: Participants
Arm/Group | Alianza Latina
Number analyzed (Participants) | 100
Participants
  Not at all | 7
  Somehow | 13
  Very | 52
  Extremely | 15
  Missing | 12
  Does not know | 1

13. Primary Outcome: Overall Participant Satisfaction With the Navigator Side of the Intervention
Description: Survey question to the caregiver including a 5-item Likert scale on satisfaction with Navigator services (not at all to very much)
Time Frame: 6 months after baseline
Population: Participants responding to these are caregivers
Measure: Count of Participants; unit: Participants
Arm/Group | Alianza Latina
Number analyzed (Participants) | 100
Participants
  Not at all | 0
  Somehow | 5
  Very | 43
  Extremely | 40
  Missing | 12

14. Primary Outcome: Participant Suggestions of Improvement
Description: Survey question to the caregiver including an open-ended question about which aspects of the intervention they would change
Time Frame: 6 months after baseline
Population: Participants responding to these are caregivers
Measure: Count of Participants; unit: Participants
Arm/Group | Alianza Latina
Number analyzed (Participants) | 100
Participants
  Responded | 88
  Missing | 12

15. Primary Outcome: Practitioner Adherence to Guideline Recommendations
Description: 10-item checklist administered to the dyads asking about the implementations of different aspects of dementia service guidelines
Time Frame: 6 months after baseline
Population: 87 respondents
Measure: Median (Inter-Quartile Range); unit: Guideline Items in the checklist covered
Arm/Group | Alianza Latina
Number analyzed (Participants) | 87
Guideline Items in the checklist covered | 9 [6 to 10]

16. Secondary Outcome: Patients' Behavioral Symptoms
Description: Brief version of the Neuropsychiatry Inventory Questionnaire: This is a validated clinical instrument for evaluating psychopathology in dementia. If any of the 12 neuropsychiatric symptoms is present, caregivers rate their loved one's severity on a three-point scale (mild-severe). For example, if the caregiver responds yes to "is the patient resistive to help from others at times, or hard to handle?", the following question would follow: "rate the severity of the symptom". An overall severity summary score is calculated by adding the severity scores of all items, ranging from 0 to 36, and higher scores mean higher severity.
Time Frame: Baseline and 6 months from baseline
Population: Participants responding to these are caregivers on behalf of care recipients
Measure: Mean (Standard Deviation); unit: Change in units on a scale
Arm/Group | Alianza Latina
Number analyzed (Participants) | 65
Change in units on a scale | 0.58 (6.93)

17. Secondary Outcome: Patients' Depression
Description: Short Geriatric Depression Scale: This scale measures depressive symptomatology, and consists of 15 yes vs no questions. Of the 15 items, 10 indicate the presence of depression when answered positively, while the rest (question numbers 1, 5, 7, 11, 13) indicate depression when answered negatively. A summary score is obtained ranging from 0 to 15, with higher scores meaning more severe depressive symptomatology.
Time Frame: Baseline and 6 months from baseline
Population: Participants responding to these are caregivers on behalf of care recipients or care recipients themselves when possible
Measure: Mean (Standard Deviation); unit: Change in units on a scale
Arm/Group | Alianza Latina
Number analyzed (Participants) | 65
Change in units on a scale | -0.71 (3.53)

18. Secondary Outcome: Patients' Quality of Life
Description: Quality of Life in Alzheimer's Disease: The Quality of Life in Alzheimer's Disease is comprised of 13 items (physical health, energy, mood, living situation, memory, family, marriage, friends, self as a whole, ability to do chores, ability to do things for fun, money and life as a whole). Response options include 1(poor), 2(fair), 3(good) and 4 (excellent), for a total score of 13-52, with higher scores indicating better quality of life.
Time Frame: Baseline and 6 months from baseline
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Change in units on a scale
Arm/Group | Alianza Latina
Number analyzed (Participants) | 65
Change in units on a scale | 0.42 (6.07)

19. Secondary Outcome: Caregivers' Quality of Life
Description: In general, how satisfied are you with your life?" with a 4-point scale from 1 (Very Satisfied) to 4 (Very Dissatisfied)
Time Frame: Baseline and 6 months from baseline
Population: Participants responding to these are caregivers on their behalf
Measure: Mean (Standard Deviation); unit: Change in units on a scale
Arm/Group | Alianza Latina
Number analyzed (Participants) | 77
Change in units on a scale | 0.14 (0.79)

20. Secondary Outcome: Caregivers' Depression
Description: 10-item Center for Epidemiologic Studies-Depression scale (CES-D-10): This is a 10-item, self-report rating scale that measures characteristic symptoms of depression in the past week (e.g. depression, loneliness, restless sleep). Each item is rated on a 4-point scale, from 0 (rarely or none of the time) to 3 (most or all of the time) with positively worded items (items 5 and 8) reverse scored. Items yield summary scores that range from 0 to 30, with higher scores indicating higher severity. An example of an item is: "I was bothered by things that usually don't bother me"
Time Frame: Baseline and 6 months from baseline
Population: Participants responding to these are caregivers on their behalf
Measure: Mean (Standard Deviation); unit: Change in units on a scale
Arm/Group | Alianza Latina
Number analyzed (Participants) | 77
Change in units on a scale | -0.43 (6.22)

21. Secondary Outcome: Caregivers' Burden
Description: Short Zarit Burden Interview: This caregiver burden scale has 6 items that address the perceived impact of the act of providing care on the physical health, emotional health, social activities and financial situation of the caregiver. Each item has five response options ranging from "never" to "nearly always". A total score is obtained by adding scores in all items, with a range from 0 to 24. Higher scores mean higher burden.
Time Frame: Baseline and 6 months from baseline
Population: Participants responding to these are caregivers on their behalf
Measure: Mean (Standard Deviation); unit: Change in units on a scale
Arm/Group | Alianza Latina
Number analyzed (Participants) | 77
Change in units on a scale | 0.34 (4.32)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse Events were not monitored in any participant population due to this project being minimal risk. instead, the research team monitored unanticipated problems.
Groups:
- Alianza Latina: The main components of Alianza Latina are 1) providing primary care providers with education, training and tools for timely dementia diagnosis and optimal treatment and 2) providing Latino dementia patients with enhanced chronic care through bilingual Health Navigators. This number includes 100 caregivers of 84 care recipients who underwent the Alianza Latina care support intervention; 26 caregivers were part of 10 clusters of 2 (n=5), 3 (n=4), and 4 (n=1) caregivers of the same person with dementia. This number also includes results from 59 primary care providers who underwent a dementia training delivered as standard training by the KU Alzheimer's Disease Research Center. Data for all 3 groups are provided together because they are part of the same intervention, and not interventions that were compared. Mortality only happened among care recipients.
Arm/Group | Alianza Latina
All-Cause Mortality (participants affected / at risk) | 6/243
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-06): https://cdn.clinicaltrials.gov/large-docs/32/NCT04418232/Prot_SAP_000.pdf
  • Informed Consent Form (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/32/NCT04418232/ICF_001.pdf